CLINICAL TRIAL: NCT03095664
Title: Effect of a Lifestyle Intervention on Nutritional Status and Prognosis of Endometrial Cancer Survivors
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped due to COVID-19 pandemic, as conducting a behaviour-change programme in groups was not recommended to prevent the spread of the virus.
Sponsor: Brazilian National Cancer Institute (Other Government)
Responsible Party: Principal Investigator, Gabriela Villaça Chaves, PhD, researcher, Brazilian National Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 55155116.9.0000.5274
Record Dates: First submitted 2017-03-14; First posted 2017-03-30 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Endometrium Cancer; Life Style; Obesity
Keywords: lifestyle intervention; endometrial cancer; survival
MeSH Terms: conditions — Endometrial Neoplasms; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): 6 months after surgical treatment, women in the experimental group will attend a counseling program to promote healthy eating and physical activity.
  Interventions: Behavioral: Intervention group
- Control group (No Intervention): Control group will receive usual care (verbal nutritional counseling after surgical treatment, at discharge).

INTERVENTIONS:
Behavioral: Intervention group — A behavior change program with 4 monthly 90-min sessions about healthy eating and physical activity.
  Other Names: Lifestyle intervention counseling program
  Arms: Intervention group

SUMMARY:
The objective of the present study is to implement and evaluate the effect of a counseling program to promote healthy eating and practice of physical activity in the nutritional status, quality of life and prognosis of women Type I (endometrioid) endometrial cancer.

DETAILED DESCRIPTION:
Endometrial cancer (EC) is the fifth most commonly diagnosed malignant neoplasm among women worldwide. The incidence of EC is higher in high-income countries, but it has been increasing in low- and middle-income countries.

The main risk factors for EC include the presence of comorbidities, such as diabetes mellitus and hypertension, as well as conditions associated with prolonged exposure to estrogens. Obesity is recognized as a major risk factor for many cancers, including EC. Multiple mechanisms related to obesity are probably involved in the carcinogenesis of EC. Among obese women in the postmenopausal period, there is an increase of bioavailable circulating estrogens. These estrogens come from the aromatization of androgens in adipose tissue and from increased circulating estrogens secondary to the reduced synthesis of sex hormone binding globulin (SHBG) in the liver. Insulin resistance, hyperinsulinemia, increased secretion of adipocytokines and pro-inflammatory cytokines may also play a role in the carcinogenesis of EC.

Although the incidence of EC is remarkable, insufficient data has addressed the impact of obesity on EC outcomes. Since about 70% of women diagnosed with endometriod EC are obese, the consequences of obesity-related diseases should be taken into account in order to implement strategies to improve survival outcomes among these women.

Sedentary lifestyle and physical inactivity also seem to be relevant, and have been identified as predictors of poor prognosis in patients with different types of cancer. However, the role of lifestyle (including eating and social habits and physical activity) on endometrial cancer prognosis has not been assessed prospectively yet. Studies assessing nutritional status and lifestyle before and after EC diagnosis may elucidate whether and when these factors influence clinical outcomes, including long-term survival.

ELIGIBILITY:
Inclusion Criteria:

* endometrial cancer patients undergoing surgical treatment

Exclusion Criteria:

* previous oncologic treatment
* cancer stage IV according to the International Federation of Gynecology and Obstetrics (FIGO)
* patients who report physical activity over 150 minutes/week of moderate or vigorous intensity
* individuals with decompensated diabetes mellitus or hypertension
* patients who have a contraindication to physical activity.

Ages: 20 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  mortality after 5 years

SECONDARY OUTCOMES:
Change in Quality of life | 0, 6, 12, 24, 26, 48 and 60 months after surgery
  Change in quality of life assessed by the Quality of Life-30 (QL30) questionaire of the European Organisation for Research and Treatment of Cancer (EORCT) before and 6, 12, 24, 26, 48 and 60 months after surgery.
Change in handgrip strength | 0, 6, 12, 24, 26, 48 and 60 months after surgery
  Change in handgrip strength before and 6, 12, 24, 26, 48 and 60 months after surgery.
Change in functional capacity (30 second stand chair test) | 0, 6, 12, 24, 26, 48 and 60 months after surgery
  change in functional capacity assessed by 30 second stand chair test before and 6, 12, 24, 26, 48 and 60 months after surgery
Change in functional capacity (Timed Get Up and Go test) | 0, 6, 12, 24, 26, 48 and 60 months after surgery
  change in functional capacity assessed by Timed Get Up and Go test before and 6, 12, 24, 26, 48 and 60 months after surgery
Change in functional capacity (6 minute walk test) | 0, 6, 12, 24, 26, 48 and 60 months after surgery
  change in functional capacity assessed by 6 minute walk test before and 6, 12, 24, 26, 48 and 60 months after surgery
Change in Physical activity behaviour | 0, 6, 12, 24, 26, 48 and 60 months after surgery
  change in physical activity behaviour assessed by The International Physical Activity Questionnaire (IPAQ) before and 6, 12, 24, 26, 48 and 60 months after surgery
Change in food intake pattern | 0, 6, 12, 24, 26, 48 and 60 months after surgery
  change in food intake pattern assessed by Food Frequency questionaire before and 6, 12, 24, 26, 48 and 60 months after surgery
Change in Body composition | 0, 6, 12, 24, 26, 48 and 60 months after surgery
  change in body composition assessed by bioelectrical impedance before and 6, 12, 24, 26, 48 and 60 months after surgery
Change in anthropometric status (weight) | 0, 6, 12, 24, 26, 48 and 60 months after surgery
  change in weight before and 6, 12, 24, 26, 48 and 60 months after surgery
Change in anthropometric status (body mass index) | 0, 6, 12, 24, 26, 48 and 60 months after surgery
  change in body mass index before and 6, 12, 24, 26, 48 and 60 months after surgery
Change in anthropometric status (waist circumference) | 0, 6, 12, 24, 26, 48 and 60 months after surgery
  change in waist circumference before and 6, 12, 24, 26, 48 and 60 months after surgery
Change in anthropometric status (hip circumference) | 0, 6, 12, 24, 26, 48 and 60 months after surgery
  change in hip circumference before and 6, 12, 24, 26, 48 and 60 months after surgery
Disease-free survival | 5 years
  Disease-free survival after 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela V Chaves, PhD, Principal Investigator — Brazilian National Cancer Institute
Locations (1):
- Brazilian National Cancer Institute, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agnew H, Kitson S, Crosbie EJ. Interventions for weight reduction in obesity to improve survival in women with endometrial cancer. Cochrane Database Syst Rev. 2023 Mar 27;3(3):CD012513. doi: 10.1002/14651858.CD012513.pub3. PMID 36971688